CLINICAL TRIAL: NCT06891001
Title: The Utilization of a Shoe Insert on Individuals With Unilateral Greater Trochanteric Pain Syndrome on Single Leg Stance, Biomechanics, and Pain Intensity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Daniel S. Cooper, Physical Therapist, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-011290
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Gluteus Medius Muscle Strength; Lateral Hip Pain; Greater Trochanter Pain Syndrome, Gluteus Medius Tendinopathy, Gluteus Minimus Tendinopathy
Keywords: Gluteus medius tendinopathy; Gluteus minimum tendinopathy; Greater trochanteric pain syndrome
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Therapy (Active Comparator): This arm will undergo a standardized physical therapy protocol alone.
  Interventions: Other: Physical Therapy
- Physical Therapy Plus Bilateral Shoe Insert (Sham Comparator): This arm will undergo a standardized physical therapy protocol with the addition of a neutral shoe insert bilaterally.
  Interventions: Device: Bilateral Shoe Insert
- Physical Therapy Plus Unilateral Shoe Insert (Experimental): This arm will undergo a standardized physical therapy protocol with the addition of a neutral shoe insert on the involved side.
  Interventions: Device: Unilateral neutral shoe insert

INTERVENTIONS:
Device: Unilateral neutral shoe insert — In the treatment group, subjects will undergo the addition of a neutral shoe insert to the involved lower extremity according to manufacturer guidelines at the initial visit. These subjects will also undergo a once-weekly 12-week course of physical therapy according to the established standardized protocol.
  Arms: Physical Therapy Plus Unilateral Shoe Insert
Device: Bilateral Shoe Insert — For subjects placed in the sham group, subjects will undergo the addition of a neutral shoe insert to both lower extremities according to manufacturer guidelines at the initial visit. These subjects will also undergo a once-weekly 12-week course of physical therapy according to the established standardized protocol with guidelines .
  Arms: Physical Therapy Plus Bilateral Shoe Insert
Other: Physical Therapy — For subjects placed in the control group, subjects will undergo a once-weekly 12-week course of physical therapy according to the established standardized protocol.
  Arms: Physical Therapy

SUMMARY:
We hypothesize that the addition of a unilateral neutral shoe insert combined with standard physical therapy (PT+SI) will have greater improvements in pain and function at 12 weeks and 6 months compared to physical therapy with sham inserts (PT+Sham) and physical therapy (PT) alone. In addition, we hypothesize that the addition of a neutral shoe insert in the involved limb will immediately improve biomechanics and pain with the single-leg stance test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of unilateral hip pain lasting more than three months.
* Subjects with a VAS pain score of at least 3/10 localized to the lateral hip.
* Subjects with pain with palpation to lateral hip.
* Subjects with pain with either resisted hip abduction in relative adduction testing position and/or single leg stance test

Exclusion Criteria:

* Subjects wearing custom foot orthoses at the time of recruitment.
* Subjects who endorse current low back pain ≥ 3 on the NRS or lumbar radiculopathy
* Subjects with a medical history of spinal or lower limb surgery in the past 6 months.
* Subjects with a medical history of total joint replacement of hip, knee, or ankle on the symptomatic side
* Subjects who have had a corticosteroid injection at the hip within the last 12 months;
* Subjects demonstrating clinical signs and symptoms of intra-articular hip joint pathology with ≥ 3/10 groin pain including imaging confirmed significant labral tearing requiring surgery or osteoarthritis > 2 (mild) on Kellgren-Lawrence score on radiographs.
* Subjects previously diagnosed with systemic inflammatory conditions; active cancer/malignant tumors; or neurological conditions that would affect gait
* Subjects who have had physical therapy within the past 3 months for hip pain
* If subjects are unable to commit to 12 weeks of therapy with one supervised session weekly
* Subjects who have the intention to perform treatments outside of this study including, but not limited to, dry needling or acupuncture, extracorporeal shockwave, therapeutic ultrasound, a TENEX procedure, medication injection therapies, platelet-rich plasma injections, stem cell injections, and surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute Sport Assessment - Gluteal Questionnaire | 12 weeks
  The VISA-G is a self-reported scale to quantify disability associated with gluteal tendinopathy. The instrument is freely available, and scores range from 0-100, with 100 indicating no hip-related disability and 0 indicating fully disabled. The questionnaire includes eight items asking questions about usual pain (item 1), pain with tendon loading (items 2, 3, 4, and 6), difficulty moving after sitting (item 5), and activity participation (items 7 and 8). Item 8 asks the subject to choose one of 3 sections (A, B, or C) and check the appropriate response related to the ability to perform weight-bearing activities including walking, shopping, or running.

SECONDARY OUTCOMES:
Visual Analog Scale for Pain | 12 weeks
  The Visual Analog Scale for Pain is a measurement instrument that is used to quantify pain and discomfort by having an individual select a number on a Likert scale between 0 and 10, with 0 being no pain and 10 being the worst imaginable pain.
Global Rating of Change Scale | 12 weeks
  The GROC scale is a single-item instrument that asks the subject to rate the global or overall change and to what extent, if any, since initiating treatment. The GROC uses a Likert scale to indicate the direction of change (worsening or improving) and to what extent ("tiny" to "very great"). This scale is only administered after treatment has occurred and is not necessary prior to initiation of treatment.
Isometric Hip Strength | 12 weeks
  The subject will be placed supine with the uninvolved knee bent/foot on the table. The affected/other leg will be straight with knee fully extended with a gait belt anchored around the table and leg. A handheld dynamometer measuring in Newtons will be in between the gait belt and leg and the sensor will be placed 5 cm proximal to the lateral malleoli. The subject will be asked to abduct/lift the leg out to the side with as much force as possible against the dynamometer for 5 seconds. Two trials will be completed.
Single Leg Stance for Pain | 12 weeks
  Subject stands on test leg/one leg with an opposite fingertip on the wall for balance for up to 30 seconds. A positive test is a familiar pain. The examiner will note the subjects' pain rating via VAS. A neutral shoe insert will be added to the subjects' stock shoe insert and the test will be repeated again noting the pain rating to assess for any changes.
Single Leg Stance Biomechanics | 12 weeks
  Prior to the test, the examiner will place a total of six reflective markers on the patient. The markers will be placed on the bilateral acromion process of the scapula, the bilateral anterior superior iliac spine, and the bilateral second metatarsal head. A first photograph will be taken of the subject in a bilateral-limb stance. The participant will be asked to balance in a single-leg stance. Once the patient is in a single-leg stance, a photo will be taken every 0.5s for 2s. A second grouping of photos will be taken with the patient standing in a single-limb stance with the addition of a neutral heel lift. Retrospective analysis will be performed on these photos. The mean values of the angles will be calculated using the analysis software. The angles to be calculated include the trunk sway angle, the pelvic tilt angle, and the pelvic-on-femur angle.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Glendale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided